CLINICAL TRIAL: NCT06592391
Title: Process Evaluation and Effectiveness Trial to Assess a Tailored Whole School Approach for a More Dynamic School Day in Dutch Primary Schools.
Brief Title: A Study on an Educational Tool for the Development of a Tailored Dynamic School Day in Dutch Primary Schools.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam University of Applied Sciences (Other)
Collaborators: Hanze University of Applied Sciences Groningen (Other); Fontys University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HVA-271
Record Dates: First submitted 2024-07-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Physical Activity; Children, Only
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- expert schools (Other): These schools developed their own dynamic school day over the past 5 - 10 years without using the educational innovation.
  Interventions: Other: expert schools
- Cohort 1 (Experimental): These schools will start the development of a tailored dynamic school day using the educational innovation in September 2024. The educational component consists of a number of face-to-face meetings. The implementation of the local plans will start September 2025.
  Interventions: Other: educational innovation dynamic school day
- Cohort 2 (Experimental): these schools will start the development of a tailored dynamic school day using the e-learning version of the educational innovation in September 2025. The implementation of the local plans will start September 2026.
  Interventions: Other: e-learning on a dynamic school day

INTERVENTIONS:
Other: educational innovation dynamic school day — Schools will form a community of practice, and will be supported with regular workshop to develop a dynamic school day that matches the local context.
  Arms: Cohort 1
Other: e-learning on a dynamic school day — Schools will form a community of practice, and will develop a dynamic school day that matches their local context using e-learning materials
  Arms: Cohort 2
Other: expert schools — Schools that have developed a local dynamic school day without additional support
  Arms: expert schools

SUMMARY:
A dynamic school day is a school day that involves regular interruptions of sedentary learning with moments of physical activity. Many Dutch primary schools have thus far not succeeded in making their school day more 'dynamic' .

In this project, the researchers will develop an educational innovation to support schools in the development of a dynamic school day that is tailored to their local context. To determine the effectiveness of the educational innovation, the researchers will study the implementation process and assess the effectiveness.

The research questions for the researcher project are:

1. To what extend are school teams successful in the development and implementation of a tailored dynamic school day, and what are facilitating and hindering factors during implementation?
2. What is the effect of the tailored dynamic school day on 8 - 12 year old pupils? Sedentary time and physical activity behavior, wellbeing and in class behavior will be assessed.

DETAILED DESCRIPTION:
Within this project, the researchers will develop an educational innovation to support Dutch primary schools in the development of a tailored dynamic school day. To asses the effectiveness we will conduct a hybrid effect- implementation trial. The researchers will therefore conduct a process evaluation and an effectiveness trial.

The research questions for the researcher project are:

1. To what extend are school teams successful in the development and implementation of a tailored dynamic school day, and what are facilitating and hindering factors during implementation?
2. What is the effect of the tailored dynamic school day on 8 - 12 year old pupils? Sedentary time and physical activity behavior, wellbeing and in class behavior will be assessed.

Study sample:

A total of 21 schools will be invited to participate in this study. Three schools have already successfully implemented a dynamic school day in their local context on their own initiative. Those schools are called 'expert schools'. The other 18 schools (6 located in Amsterdam, 6 located in Eindhoven, 6 located in Groningen) have not structurally implemented a dynamic school day. These 18 schools will be divided over 2 cohorts that will start developing their tailored dynamic school day over the course of the project.

Cohort 1 (12 schools, evenly divided over the 3 regions) will start in September 2024 with an educational program that will support them during the development of a tailored dynamic school day. They will use a full school year to develop an implementation plan, and will start the implementation of their tailored dynamic school day from September 2025 onwards. The results of the process evaluation and effectiveness trial will be used to improve the educational innovation and develop an e-learning module.

Cohort 2 (6 schools, evenly divided over the 3 regions) will start in September 2025 with the development of their tailored dynamic school day using the e-learning module. They will also use a full school year to develop an implementation plan and start implementing from September 2026 onwards.

The process evaluation and effect assessment will be conducted in all participating schools. In the development year, a baseline measurement will be conducted in autumn. All other measurements, including the baseline measurement for the expert schools, will be conducted in the spring of each year.

ELIGIBILITY:
Inclusion Criteria:

From participating 21 schools:

* all teachers
* a board member
* all pupils from grade 4 - 8 (Dutch system, age 8 - 12)

Exclusion Criteria:

-

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 980 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
process evaluation - questionnaire | During the year of development (1st year of participation) 2 times (fall + spring school year). After that once a year (spring school year) until the end of the study which may be 2 or 3 years depending on the cohort.
  Questionnaire on experiences with the implementation of the dynamic school day
Process evaluation - semi structured interview | 1 time per year until the end of the study (spring school year) which is 2 or 3 years depending on the cohort
  Semi structured interview on school policy focussed on aspects that are related to a dynamic school day
Process evaluation - observations within the school | During the year of development (1st year of participation) 2 times (fall + spring school year). After that once a year (spring school year) until the end of the study which may be 2 or 3 years depending on the cohort.
  Observations within 2 classrooms to assess physical activity behavior during the school day
Process evaluation - analysis of teaching schedules | During the year of development (1st year of participation) 2 times (fall + spring school year). After that once a year (spring school year) until the end of the study which may be 2 or 3 years depending on the cohort.
  Teacher schedules and overview of minutes of physical activity during the schoolday to assess how many active minutes are reached.

SECONDARY OUTCOMES:
effect evaluation - wellbeing pupils | During the year of development (1st year of participation) 2 times (fall + spring school year). After that once a year (spring school year) until the end of the study which may be 2 or 3 years depending on the cohort.
  wellbeing questionnaire completed by parent of 8-12 year old pupils
effect evaluation - on-task behavior | During the year of development (1st year of participation) 2 times (fall + spring school year). After that once a year (spring school year) until the end of the study which may be 2 or 3 years depending on the cohort.
  observation within two class rooms to count the number of pupils that show on-task behavior (measured on Tuesday and Thursday)
effect evaluation - physical activity behavior | During the year of development (1st year of participation) 2 weeks (fall + spring school year). After that one week per year (spring school year) until the end of the study which may be 2 or 3 years depending on the cohort.
  Pupils will wear an accelerometer on their hip during 5 days: Monday morning - Friday afternoon